CLINICAL TRIAL: NCT04777591
Title: Effectiveness of Exparel TAP Block in Breast Free Flap Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, John Stranix, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSR210033
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain; Breast Reconstruction
Keywords: TAP block; Regional block; ERAS; liposomal bupivacaine; free flap
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Control group: TAP block with plain bupivacaine Intervention group: TAP block with plain bupivacaine + liposomal bupivacaine
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control - plain bupivacaine (Active Comparator): Receives plain bupivacaine TAP block as part of multi-modal pain control intraoperatively
  Interventions: Drug: Bupivacain
- Experimental - Liposomal bupivacaine (Experimental): Receives plain bupivacaine + liposomal bupivacaine TAP block as part of multi-modal pain control intraoperatively
  Interventions: Drug: Liposomal bupivacaine TAP block

INTERVENTIONS:
Drug: Liposomal bupivacaine TAP block — Group will receive Liposomal bupivacaine TAP block (mixed with plain bupivacaine) intraoperatively during free flap breast reconstruction as part of the multimodal pain control.
  Arms: Experimental - Liposomal bupivacaine
Drug: Bupivacain — Group will receive plain bupivacaine TAP block intraoperatively during free flap breast reconstruction as part of the multimodal pain control.
  Arms: Control - plain bupivacaine

SUMMARY:
Transversus Abdominis Plane (TAP) block is a useful tool in pain management after abdominal surgery. It is a regional nerve block that targets T6-L1 thoracolumbar nerves running in the plane between internal oblique and transversus abdominis muscle. It is shown to help with post-operative pain management, reducing pain scores and narcotic pain medication use, as well as promoting earlier return to activity and recovery. TAP block became a very popular, safe, and effective therapeutic adjunct for many different abdominal surgeries ranging from obstetric procedures to general surgery procedures like colorectal surgery. Furthermore, it is used in plastic surgery procedures such as Deep Inferior Epigastric Perforator (DIEP) free flap or Transverse Rectus Abdominis Myocutaneous (TRAM) flap, as they involve extensive amount of abdominal soft tissue incision. Previous studies have shown that TAP block in these procedures significantly reduce post-op pain and narcotic pain medication use. More recently, Exparel (liposomal bupivacaine) has risen to spotlight for providing a longer, sustained local anesthesia. Various surgical disciplines have adopted this agent as part of their pain management protocol. However, there are no literatures that describe the effect of TAP block using Exparel for breast free flap population. The study hypothesize that delivering TAP block with Exparel (vs. plain bupivacaine) will provide longer regional blocking effect, hence aiding in pain control and recovery postoperatively. The investigators will be analyzing postop narcotic pain medication requirement and pain scores to look into this question.

ELIGIBILITY:
Inclusion Criteria:

* All female patients who are 18 years or older who will undergo unilateral or bilateral abdomen-based free flap breast reconstruction at UVA Medical Center

Exclusion Criteria:

* Subjects with ages <18 years

  * Allergy to local anesthetic
  * Inability to tolerate standard postoperative pain management regimen (Tylenol, Toradol, and Oxycodone PRN) for any reason
  * Subjects who cannot read or understand English
  * Subjects who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 117 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Stranix, MD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia Medical Center, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park RH, Chou J, DeVito RG, Elmer A, Hollenbeck ST, Campbell CA, Stranix JT. Effectiveness of Liposomal Bupivacaine Transversus Abdominis Plane Block in DIEP Flap Breast Reconstruction: A Randomized Controlled Trial. Plast Reconstr Surg. 2024 Oct 1;154(4S):52S-59S. doi: 10.1097/PRS.0000000000011326. Epub 2024 Sep 20. PMID 38315156

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control - Plain Bupivacaine | Experimental - Liposomal Bupivacaine
Started | 59 | 58
Completed | 59 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Plain Bupivacaine | Experimental - Liposomal Bupivacaine | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (10.5) | 51.1 (8.7) | 51.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 58 | 117
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post-op Pain Scores During Initial Hospitalization
Description: Visual analog pain scale. Scores range from 0 to 10, 0 being no pain and 10 being worse pain that one experienced in their lifetime.
Time Frame: During initial hospitalization following surgery up to Day 5 (or to the point of discharge), whichever came first
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control - Plain Bupivacaine | Experimental - Liposomal Bupivacaine
Number analyzed (Participants) | 59 | 58
score on a scale | 4.3 [2.7 to 5.7] | 3.3 [2.2 to 5.0]

2. Primary Outcome: Post-op Narcotic Pain Medication Use During Hospitalization
Description: total amount of morphine milliequivalent
Time Frame: during initial hospitalization following surgery up to Day 5 (or to the point of discharge), whichever came first
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Control - Plain Bupivacaine | Experimental - Liposomal Bupivacaine
Number analyzed (Participants) | 59 | 58
MME | 55 [30 to 89.5] | 50 [20 to 90]

3. Secondary Outcome: Length of Hospital Stay
Description: hospital length of stay
Time Frame: during initial hospitalization following surgery up to Day 5 (or to the point of discharge), whichever came first
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control - Plain Bupivacaine | Experimental - Liposomal Bupivacaine
Number analyzed (Participants) | 59 | 58
Days | 2.1 (0.4) | 2.2 (0.6)

ADVERSE EVENTS:
Time Frame: 21 months
Arm/Group | Control - Plain Bupivacaine | Experimental - Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58
Other Adverse Events (participants affected / at risk) | 0/59 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT04777591/Prot_SAP_000.pdf